CLINICAL TRIAL: NCT00648830
Title: Randomized Single Dose Crossover Replicate Comparative Bioavailability Study of Clarithromycin 250 mg Tablets in Healthy Male and Female Volunteers Under Fasted Conditions
Brief Title: Comparative Bioavailability Study of Clarithromycin 250 mg Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mylan Pharmaceuticals Inc (Industry)
Collaborators: Genpharm ULC (Industry)
Responsible Party: Elliot Offman, Director, Biopharmaceutics, Genpharm ULC
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CAI-P4-057
Record Dates: First submitted 2008-03-31; First posted 2008-04-01 (Estimated); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Healthy
MeSH Terms: interventions — Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Clarithromycin 250 mg immediate-release oral tablet
  Interventions: Drug: Clarithromycin
- 2 (Active Comparator): Biaxin® (Clarithromycin) 250 mg tablet
  Interventions: Procedure: Clarithromycin

INTERVENTIONS:
Procedure: Clarithromycin — Single-dose of Clarithromycin 250 mg oral immediate-release tablets
  Other Names: Biaxin®, Biaxin® Filmtabs
  Arms: 2
Drug: Clarithromycin — single-dose 250 mg immediate-release oral tablets
  Arms: 1

SUMMARY:
The objective of this study was to investigate the bioequivalence of Genpharm's clarithromycin tablets following a single, oral 250 mg (1 x 250 mg) dose compared to the Biaxin® filmtab® (Abbott Laboratories USA) administered under fasted conditions. Thirty-four (34) healthy, light-, non- or ex-smoking subjects of at least 18 a years of age were randomized, in this four-period, two-treatment crossover bioequivalence study conducted by Eric Sicard, M.D. at Algorithme Pharma Inc. Montreal, Canada.

Statistical analysis of the data reveals that 90% confidence intervals are within the acceptable bioequivalent range of 80% and 125% for the natural log transformed parameters AUCT, AUCI and Cmax. This study demonstrates that Genpharm's clarithromycin 250 mg tablets are bioequivalent to Biaxin® filmtab® 250 mg tablets (Abbott Laboratories USA) administered under fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

Subjects meeting all of the following criteria may be included in the study:

Availability of volunteer for the entire study period and willingness to adhere to protocol requirements as evidenced by the informed consent form (ICF) duly signed by the volunteer

Males or females aged of at least 18 years with a body mass index (BMI) greater or equal to 19 and below 30 kg/m2

Clinical laboratory values within the laboratory's stated normal range; if not within this range, they must be without any clinical significance (laboratory tests are presented in section 6.1.1.3)

Healthy according to the laboratory results and physical examination

Light , non or ex smokers. Light smokers are defined as someone smoking 10 cigarettes or less per day, and ex smokers are defined as someone who completely stopped smoking for at least 3 months

Exclusion Criteria:

Significant history of hypersensitivity to clarithromycin, erythromycin, other macrolide antibacterial agents or any related products as well as severe hypersensitivity reactions (like angioedema) to any drugs

Presence or history of significant gastrointestinal, liver or kidney disease, or any other conditions known to interfere with the absorption, distribution, metabolism or excretion of drugs or known to potentiate or predispose to undesired effects

Presence or history of significant cardiovascular, pulmonary, hematologic, neurologic, psychiatric, endocrine, immunologic or dermatologic disease

Presence of significant heart disease or disorder according to ECG

Females who are pregnant, lactating or are likely to become pregnant during the study

Females of childbearing potential or females taking systemic contraceptives who refuse to use one of the acceptable contraceptive regimen (described in section 5.4.9) throughout the study

Positive HCG beta serum pregnancy test before or during the study

Maintenance therapy with any drug, or significant history of drug dependency or alcohol abuse (> 3 units of alcohol per day, intake of excessive alcohol, acute or chronic)

Any clinically significant illness in the previous 28 days before day 1 of this study

Use of enzyme-modifying drugs in the previous 28 days before day 1 of this study (all barbiturates, corticosteroids, phenylhydantoins, etc.)

Participation in another clinical trial in the previous 28 days before day 1 of this study

Donation of 500 mL or more of blood (Canadian Blood Services, Hema-Quebec, clinical studies, etc.) in the previous 56 days before day 1 of this study

Positive urine screening of drugs of abuse (drugs listing is presented in section 6.1.1.4)

Positive results to HIV, HBsAg or anti-HCV tests

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2004-05; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters (AUC & Cmax) | within 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sicard, M.D., Principal Investigator — Algorithme Pharma Inc
Locations (1):
- Algorithme Pharma, Montreal, Quebec, Canada

REFERENCES:
- See also: Mylan Pharmaceuticals Inc. - Clinical Trial Results — http://www.mpibiostudies.com
- See also: Daily Med - posting of most recent submitted labelling to the Food and Drug Administration (FDA) and currently in use — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Recalls, Market Withdrawals and Safety Alerts — http://www.fda.gov/opacom/7alerts.html